CLINICAL TRIAL: NCT07332806
Title: Impact of Site of Tracheal Extubation on Operating Room Efficiency During Robot-assisted Surgery: a Randomized Trial
Brief Title: Site of Tracheal Extubation and Operating Room Efficiency During Robot-assisted Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Chief Physician, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025R0568
Record Dates: First submitted 2025-12-15; First posted 2026-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Robotic Surgical Procedures; Airway Extubation; Operating Rooms; Anesthesia Recovery Period; Postoperative Complications
Keywords: Robotic Surgical Procedures; Airway Extubation; Operating Rooms; Anesthesia Recovery Period; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Airway Extubation; Operating Rooms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extubation in post-anesthesia care unit (PACU) (Experimental): At the end of surgery, patients will be transferred from operating room (OR) to PACU with endotracheal intubation and then extubated in PACU.
  Interventions: Procedure: Extubation in post-anesthesia care unit (PACU)
- Extubation in operating room (OR) (Active Comparator): At the end of surgery, patients will be extubated in operating room (OR) and then transfered to PACU.
  Interventions: Procedure: Extubation in operating room (OR)

INTERVENTIONS:
Procedure: Extubation in post-anesthesia care unit (PACU) — At the end of surgery, patients will be transfered from OR to PACU with endotracheal intubation and then extubated in PACU.
  Other Names: PACU extubation
  Arms: Extubation in post-anesthesia care unit (PACU)
Procedure: Extubation in operating room (OR) — At the end of surgery, patients will be extubated in OR and then transfered from OR to PACU.
  Other Names: OR extubation
  Arms: Extubation in operating room (OR)

SUMMARY:
This study aims to evaluate the impact of different extubation strategy on the occupancy time of operating room (OR) and the incidence of adverse events and quality of recovery after robotic-assisted surgery. The investigators hypothesize that extubation in the post-anesthesia care unit (PACU) may reduce OR occupancy time without increasing adverse events or worsening quality of recovery early after robotic-assisted surgery. This strategy may enhance perioperative efficiency while maintaining clinical safety.

DETAILED DESCRIPTION:
Major surgeries are generally performed under general anesthesia with endotracheal tube. Intubation during anesthesia induction and extubation during anesthesia emergence are two high-risk periods associated with anesthesia-related complications. In clinical practice, extubation is performed either in the OR or in the PACU, according to local routine.

Robotic-assisted surgery offers potential clinical benefits but involves high costs and limited resource availability, making operating room (OR) efficiency a critical priority. While extubation in the post-anesthesia care unit (PACU) has been suggested to improve OR turnover, evidence regarding its impact on perioperative efficiency and safety compared to standard OR extubation in robotic surgery is limited.

The investigators hypothesize that extubation in the post-anesthesia care unit (PACU) may reduce OR occupancy time without increasing adverse events or worsening quality of recovery early after robotic-assisted surgery. This study aims to evaluate the impact of different extubation strategy on the occupancy time of operating room (OR) and the incidence of adverse events and quality of recovery after robotic-assisted surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Scheduled to undergo elective robot-assisted laparoscopic surgery under general anesthesia;
3. Expected tracheal extubation during daytime working hours (before 4:00 PM).

Exclusion Criteria:

1. Refuse to participate in the study;
2. Morbid obesity (body mass index ≥35 kg/m²);
3. Preoperatively diagnosed obstructive sleep apnea, or patients with a STOP-Bang score ≥3 in combination with serum bicarbonate (HCO₃-) ≥28 mmol/L;
4. Patients at high risk of difficult airway (anticipated difficult intubation and/or extubation during preoperative assessment);
5. Preexisting sick sinus syndrome, severe sinus bradycardia (heart rate < 50 beats/min), or second-degree or higher atrioventricular block without pacemaker implantation; congenital heart disease with any type of arrhythmia; or other severe cardiovascular diseases with New York Heart Association (NYHA) functional class ≥III;
6. Significant pulmonary function impairment (FEV₁/FVC ratio < 70%, and total lung capacity [TLC] and vital capacity [VC] < 80% of predicted values);
7. Severe hepatic dysfunction (Child-Pugh class C); severe renal dysfunction (estimated glomerular filtration rate < 30 mL/min/1.73 m²); or American Society of Anesthesiologists (ASA) physical status classification ≥IV;
8. Preoperative diagnoses of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis;
9. Inability to communicate due to coma, severe dementia, or language impairment;
10. Planned postoperative admission to the intensive care unit;
11. Any other conditions that are deemed for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Operating room (OR) occupancy time | Up to 2 hours after surgery
  Time interval from end of surgery to leaving OR for PACU.

SECONDARY OUTCOMES:
Incidence of emergence delirium | Up to 3 hours after surgery
  Emergence delirium will be assessed with the confusion assessment method for the intensive care unit (CAM-ICU).
Incidence of adverse events before leaving PACU | Up to 3 hours after surgery
  An adverse event indicates any unpredictable, unfavourable medical event that is associated with any medical intervention and occurs from end of surgery to the timepoint of leaving PACU.
Time interval from end of surgery to modified Aldrete score of ≥9 | Up to 3 hours after surgery
  Modified Aldrete Score is used to assess post-anesthesia recovery in five aspects (activity, respiration, circulation, consciousness, and oxygenation); scores range from 0 to 10, with higher scores indicating better recovery. A score of ≥9 indicates that patients can be safely transferred from PACU to general wards.
Time interval from end of surgery to PACU discharge | Up to 2 hours after surgery
  Time interval from end of surgery to PACU discharge.

OTHER OUTCOMES:
Time interval from end of surgery to extubation | Up to 3 hours after surgery
  Time interval from end of surgery to extubation.
Turnover time in the operating room | Up to 3 hours after surgery
  Time interval between leaving OR of the last patient and entering OR of the next patient.
Ready for surgery time in the operating room | Up to 3 hours after surgery
  Time interval between end of surgry of the last patient and ready for surgery of the next patient.
Quality of recovery on postoperative day 1 | At 24 hours after surgery
  Quality of recovery (QoR) will be assessed using the QoR-15. QoR-15 is a 15-item scale that assesses quality of postoperative recovery in 5 domains including pain, physical comfort, physiological independence, psychological state, and support and communication. Scores range from 0 to 150, with higher scores indicating better recovery.
Length of hospital stay (LOS) after surgery | Up to 30 days after surgery
  Length of hospital stay (LOS) after surgery.
30-day all-cause mortality | Up to 30 days after surgery
  30-day all-cause mortality
Incidence of postoperative complications within 30 days | Up to 30 days after surgery
  Postoperative complications indicate any new-onset medical events that are deemed harmful and require therateutic intervention, i.e., grade 2 or higher on the Clavien-Dindo classification (grades range from I to V, with higher grade indicating more severe complications).
Total costs during hospitalization | Up to 30 days after surgery.
  Total costs during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University Fist Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godet T, Wajew C, Fabrizi M, Monet C, Pouzeratte Y, Lapeyre M, Adelou S, Pereira B, Garnier M, Chanques G, Jabaudon M, Futier E, Jaber S, De Jong A. Impact of tracheal extubation location after surgical procedures on peri-operative times: a prospective dual-centre observational study. Anaesthesia. 2025 Aug;80(8):915-926. doi: 10.1111/anae.16620. Epub 2025 May 12. PMID 40351134
- [Background] Langeron O, Bourgain JL, Francon D, Amour J, Baillard C, Bouroche G, Chollet Rivier M, Lenfant F, Plaud B, Schoettker P, Fletcher D, Velly L, Nouette-Gaulain K. Difficult intubation and extubation in adult anaesthesia. Anaesth Crit Care Pain Med. 2018 Dec;37(6):639-651. doi: 10.1016/j.accpm.2018.03.013. Epub 2018 May 23. PMID 29802903
- [Background] Thilen SR, Weigel WA, Todd MM, Dutton RP, Lien CA, Grant SA, Szokol JW, Eriksson LI, Yaster M, Grant MD, Agarkar M, Marbella AM, Blanck JF, Domino KB. 2023 American Society of Anesthesiologists Practice Guidelines for Monitoring and Antagonism of Neuromuscular Blockade: A Report by the American Society of Anesthesiologists Task Force on Neuromuscular Blockade. Anesthesiology. 2023 Jan 1;138(1):13-41. doi: 10.1097/ALN.0000000000004379. PMID 36520073
- [Background] Apfelbaum JL, Hagberg CA, Connis RT, Abdelmalak BB, Agarkar M, Dutton RP, Fiadjoe JE, Greif R, Klock PA, Mercier D, Myatra SN, O'Sullivan EP, Rosenblatt WH, Sorbello M, Tung A. 2022 American Society of Anesthesiologists Practice Guidelines for Management of the Difficult Airway. Anesthesiology. 2022 Jan 1;136(1):31-81. doi: 10.1097/ALN.0000000000004002. PMID 34762729
- [Background] Banik RK, Honeyfield K, Qureshi S, Reddy SG. Incidence and Mortality Rate of Perioperative Reintubation: Case Series of 196 Patients. AANA J. 2021 Dec;89(6):476-479. PMID 34809752
- [Background] Chen S, Zhang Y, Che L, Shen L, Huang Y. Risk factors for unplanned reintubation caused by acute airway compromise after general anesthesia: a case-control study. BMC Anesthesiol. 2021 Jan 12;21(1):17. doi: 10.1186/s12871-021-01238-4. PMID 33435881
- [Background] Koga K, Asai T, Vaughan RS, Latto IP. Respiratory complications associated with tracheal extubation. Timing of tracheal extubation and use of the laryngeal mask during emergence from anaesthesia. Anaesthesia. 1998 Jun;53(6):540-4. doi: 10.1046/j.1365-2044.1998.00397.x. PMID 9709138